CLINICAL TRIAL: NCT00616070
Title: Study of Difluprednate in the Treatment of Inflammation Following Ocular Surgery (ST-601-003)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sirion Therapeutics, Inc. (Industry)
Responsible Party: Roger Vogel, MD, Sirion Therapeutics
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST-601-003
Record Dates: First submitted 2008-02-04; First posted 2008-02-15 (Estimated); Last update posted 2011-06-30 (Estimated); Status verified 2011-06

CONDITIONS: Inflammation
MeSH Terms: conditions — Inflammation | interventions — difluprednate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental): Difluprednate
  Interventions: Drug: Difluprednate
- 2 (Placebo Comparator): Vehicle
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Difluprednate — Difluprednate
  Arms: 1
Other: Placebo — Vehicle
  Arms: 2

SUMMARY:
The purpose of this phase III study is to determine the safety and efficacy of difluprednate in the management of inflammation following ocular surgery.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for unilateral ocular surgery.

Exclusion Criteria:

* Systemic administration of any corticosteroid or immunosuppressive drug in the 2 weeks prior to study enrollment.

Min Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
The proportion of subjects with an anterior chamber cell grade of "0" and a flare grade of "0" on Day 14, compared between difluprednate and placebo groups | Day 14

SECONDARY OUTCOMES:
The proportion of subjects with an anterior chamber cell grade of "0" and a flare grade of "0" on Day 7, compared between difluprednate and placebo groups. | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Roger Vogel, MD, Study Chair — Sirion Therapeutics
Locations (1):
- Charlotte Eye, Ear, Nose & Throat, Charlotte, North Carolina, United States